CLINICAL TRIAL: NCT00180063
Title: Characterization of Local Vascular Effects of LNMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IKPD 01-02 Amend LNMMA
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-11-02 (Estimated); Status verified 2005-09

CONDITIONS: Healthy Subjects

INTERVENTIONS:
Drug: L-NMMA(drug)

SUMMARY:
Characterization of an unexpected venodilative effect of higher L-NMMA-doses in dorsal human hand veins.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* any relevant disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2003-10; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Kirch, MD, Study Chair — Institute of Clinical Pharmacology
Locations (1):
- Institute of Clinical Pharmacology, Medical Faculty, University of Technology, Dresden, Germany

REFERENCES:
- [Derived] Schindler C, Leuschner S, Schwanebeck U, Kirch W. Characterization of local vascular effects of the nitric oxide inhibitor NG-monomethyl-L-arginine on dorsal hand veins. J Clin Pharmacol. 2012 Jun;52(6):859-69. doi: 10.1177/0091270011406277. Epub 2011 May 12. PMID 21566204